CLINICAL TRIAL: NCT01452308
Title: A Phase 2a, Pilot, Open-Label Trial Evaluating the Safety, Tolerability and Pharmacodynamic Effects of GS-6624 in Subjects With Fibrosis of the Liver
Brief Title: Pilot Study of Simtuzumab in the Treatment of Liver Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-321-0101
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Liver Fibrosis
Keywords: Gilead; Gilead Sciences; GSI; Liver Fibrosis; Liver; Fibrosis
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis | interventions — simtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Participants will receive simtuzumab at a dose of 10 mg/kg by intravenous (IV) infusion every other week for a total of 3 infusions.
  Interventions: Biological: Simtuzumab
- Cohort 2 (Experimental): Participants will receive simtuzumab IV every other week for a total of 3 infusions. The dose will depend on the safety and tolerability of simtuzumab seen in Cohort 1 but will not exceed 20 mg/kg.
  Interventions: Biological: Simtuzumab

INTERVENTIONS:
Biological: Simtuzumab
  Other Names: GS-6624

SUMMARY:
This study will evaluate the safety and tolerability of simtuzumab (GS-6624) in patients with fibrosis of the liver.

Up to 20 participants will be enrolled into two sequential cohorts. Cohort 1 will consist of 10 participants who will receive simtuzumab every other week for a total of 3 infusions. Participants in Cohort 2 (10 subjects) will also receive simtuzumab every other week for a total of 3 infusions; the dose will depend on the safety and tolerability of simtuzumab seen in Cohort 1.

Participants from both cohorts who have completed the main study will be allowed to continue on simtuzumab treatment for an additional extension period, and will receive up to 13 additional infusions of simtuzumab at a fixed dose of 700 mg for an additional 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 - 65 years of age
* Chronic liver disease of any etiology
* Stage 1-3 fibrosis by Metavir score on a liver biopsy.
* Body mass index <36 kg/m2

Exclusion Criteria:

* Any evidence of hepatic decompensation past or present
* Subjects currently abusing amphetamines, cocaine, opiates, or alcohol
* Clinically significant cardiac disease
* History of cancer, other than non-melanomatous skin cancer, within 5 years prior to Screening
* Systemic fungal, bacterial, viral, or other infection that is not controlled
* Use of systemic immunosuppressants within 28 days of the Pre-treatment Phase
* Use of approved therapy for hepatitis C or hepatitis B virus within 28 days of the Pre-treatment Phase
* Pregnant or lactating
* History of bleeding diathesis within the last 6 months of study Day 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events on multiple, escalating IV doses of simtuzumab | Through Week 14
  The endpoints to be evaluated will include graded Adverse Events, laboratory abnormalities, and vital sign measurements

SECONDARY OUTCOMES:
Assessment of serum concentration of simtuzumab | Through Week 14
  Trough concentrations will be summarized by day, treatment and dose.
Antibody formation to simtuzumab (anti-simtuzumab Abs) | Through Week 14
  Immunogenicity endpoints will be geometric mean titer (GMT) and geometric mean fold rate (GMFR) for a select set of antibodies.
Measurement of pharmacodynamic (PD) markers after administration of simtuzumab | Through Week 14
  Pharmacodynamic markers include: Tissue PD markers through mRNA expression, LOXL2, LOX, Other LOXL proteins, αSMA, Collagen 1A1, NFKB1, Caspase 1, SMAD, and NOD; Serum and plasma PD markers include: APRI, LOXL2, Osteopontin, Hyaluronic Acid, CXCL 9, 10 and 11, MMP1, MMP3, MMP9, TIMP1, CD40L, TGF-β1, ET-1, VEGF, GAL3, IL-6 / IL-8 / TNFα / IFNγ, α2-macroglobulin, Apolipoprotein A1.
Assessing the effects of chronic dosing of simtuzumab on liver structure and fibrotic markers | Up to 24 weeks
  Measuring the effect of an additional 24 weeks of simtuzumab dosing on liver histology, LOXL2 and mRNA expression in the liver and serum markers of liver fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Bornstein, MD, Study Director — Gilead Sciences
Locations (1):
- Weill Cornell Medical College: NewYork-Presbyterian Hospital, New York, New York, United States